CLINICAL TRIAL: NCT01586351
Title: Arthroscopic Rotator Cuff Reconstruction With Xenologous Dermis-patch Augmentation and ACP® - Injection in Patients Over 60 Years (ACP = Autologous Conditioned Plasma)
Brief Title: Rotator Cuff Reconstruction With Xenologous Dermis-patch Augmentation and ACP® - Injection
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Principal Investigator, Matthias Flury, Principal Investigator (Department of Upper Extremity), Schulthess Klinik
Other Study IDs: ACP02
Record Dates: First submitted 2012-04-24; First posted 2012-04-26 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff tears; ACP; DX Reinforcement Matrix
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patch and ACP Treatment: Patents who get an patch augmentation and ACP injection following an arthroscopic repair of the rotator cuff.
  Interventions: Device: Patch Augmentation and ACP injection

INTERVENTIONS:
Device: Patch Augmentation and ACP injection — Patch augmentation and 4mL autologous conditioned plasma application under the footprint following an arthroscopic repair of the rotator cuff.
  Other Names: ACP; DX Reinforcement Matrix

SUMMARY:
The purpose of this study is to show that an augmentation with the DX Reinforcement Matrix from Arthrex is possible with the arthroscopic technique.

DETAILED DESCRIPTION:
The shoulder joint, specially the rotator cuff, is one of the most complicated joints of the human body. If the tendon has to be fixed at the bone during surgery, the weak point in obtaining a successful surgery is the fixation of the tendon at the bone insertion site. Tendon belongs to the bradytrophic tissue conditional on the reduced blood flow, deep mitosis rate and lowered healing potential.

The patients in this study have 60 years or more. The tissue of these patients isn't as good as in young patients. The patch will be used to improve the strength of the tendon at the insertion site and the ingrowth process of the new tissue at this area. Additionally the investigators can boost the healing process with a selective use of PRP (PRP = platelet rich plasma). In this process, the healing site is delivered with an elevated concentration of thrombocytes and also growth factors which are constituent parts of them.

ELIGIBILITY:
Inclusion Criteria:

* Arthroscopic rotator cuff reconstructions of degenerative or traumatic full thickness rotatorcuff tears (supraspinatus should be affected)performed by Dr. Flury
* Age: 60 years or more
* Suture bridge technique
* Women: No longer of childbearing age (at menopause and last menstrual period more than 12 months, prevented surgically Ovaries and/or uterus removed surgically)
* Signed consent form

Exclusion Criteria:

* Partial reconstruction of the rotator cuff (PASTA)
* Open reconstruction
* Tendon transfer (latissimus dorsi or pectoralis major)
* Revision surgery
* Omarthrosis (Level ≥ 2 Samilson & Prieto)
* Systemic arthritis
* Rheumatoid arthritis
* Diabetes (insulin treated)
* Requiring surgery in reconstruction of the subscapularis tendon
* Progressive fat inclusion (fatty infiltration of the rotator cuff musculature goutallier level IV
* Acute or chronic infection
* Pathological bone metabolism
* Insufficient perfusion in the affected arm
* Neuromuscular disease in the affected arm
* Non compliance of the patient
* Disorders which handicap or inhibit the patient to follow the orders of the clinical testers

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The potential patients will be recruited from the operation list due to the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Oxford Shoulder Score (Questionnaire) | 3mo
  The Oxford Shoulder Score used after 3 months is the primary parameter. The Score tests the ability to participate in the patients' normal life before they got injured.

SECONDARY OUTCOMES:
VAS Pain Scoring Tool | 10d
  Measuring of the pain with a VAS pain scale during 10 days post-operative
QuickDASH Questionnaire (Short version of Disability of the Arm, Shoulder and Hand Questionnaire) | 3/6/24mo
  The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb.
  The QuickDASH is a shortened version of the DASH Outcome Measure. Instead of 30 items, the QuickDASH uses 11 items to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb.
EQ-5D Questionnaire | 3/6/24 mo
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal.Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys.
ROM (degrees) | 3/6/24mo
  Range of motion refers to the distance and direction a joint can move.
Measurement of the abduction strength (Kilograms) | 3/6/24 mo
ASES Score (American Shoulder And Elbow Surgeons Questionnaire) | 3/6/24mo
  The ASES was developed to measure functional limitations and shoulder pain in people with musculoskeletal pathologies. Pain score was calculated from a single pain question on a visual analog scale (pain symptoms) and a function score from the sum of 10 questions addressing function using a 4-point ordinal scale (physical function). Pain and function are weighted equally and the total score ranges from 0 to 100 points, where 0 = worst and 100 = best.
Constant Murley Score (CMS) | 3/6/24 mo
  The CMS is a 100-point scoring system that is divided into four subscales: pain (15 points), activities of daily living (20 points), range of motion (40 points) and strength (25 points).Pain and activities of daily living are self-reported by the patient using visual analog scales and ordinal categories. Range of motion is obtained during active painfree elevation in flexion and abduction (using a goniometer), and functional internal and external rotation of the shoulder (using ordinal scale). Strength testing was performed at 90° of abduction in the scapular plane.
MRI/X-Ray/Ultrasonic Diagnostics (Objective Evaluation (Descriptive) of the healing process) | 6/24 mo
Measurement of the external rotation strength (Kilograms) | 3/6/24 mo
Oxford Shoulder Score (Questionnaire) | 6mo/24mo
  The Oxford Shoulder Score used after 3 months is the primary parameter. The Score tests the ability to participate in the patients' normal life before they got injured.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Flury, Dr, Principal Investigator — Upper Extremities Department
Locations (1):
- Schulthess Klinik, Zurich, Canton Zürich, Switzerland